CLINICAL TRIAL: NCT01790282
Title: Is E2 Luteal Support in High Responder Long Gn-RH Agonist ICSI Cycles Detrimental to Cycle Outcome ? A Randomized Clinical Trial
Brief Title: Is Adding E2 to P4 Luteal Support In High Responder Long Gn-RH Agonist ICSI Cycles Detrimental to Outcome? RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura Integrated Fertility Center (Other)
Responsible Party: Principal Investigator, Emad Mohamad Sedeek, Dr, Mansoura Integrated Fertility Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2 luteal support in ICSI
Record Dates: First submitted 2013-02-08; First posted 2013-02-13 (Estimated); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: IVF; Infertility
Keywords: luteal support; high responder; ICSI; cycle outcome
MeSH Terms: conditions — Infertility | interventions — Estradiol; Progesterone; Injections, Intramuscular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- estradiole - progesterone arm (Experimental): Cases are given estradiole valerate 2mg 3 times /day from day of ovum pick up until the time of pregnancy test two weeks together with daily IM injection of 100 progesterone starting . Single intramuscular 0.1 mg decapeptyl are given on day of transfer
  Interventions: Drug: estradiol plus progesterone 100 mg IM injection; Drug: Progesterone IM of 100 mg
- Progesterone only arm (Active Comparator): Patient are given 100 mg progesterone daily starting on day of pickup plus single dose of decapeptyl 0.1 mg on day of embryo transfer
  Interventions: Drug: Progesterone IM of 100 mg

INTERVENTIONS:
Drug: estradiol plus progesterone 100 mg IM injection — estradile valaerate 2mg plus progesterone 100 mg/day support arm :E2 valerate 2mg three times /day are given to the arm cases plus P4 100 IM/day for 14 days starting on day of ovum pickup and single IM injection of 0.1 mg decapeptyl on day of ET
  Other Names: estradiole valerate 2mg,; Prontogest 100 mg
  Arms: estradiole - progesterone arm
Drug: Progesterone IM of 100 mg — Starting on day of ovum pickup ICSI cases are given prontogest 100 mg IM /day plus single dose dose of treptorline 0.1mg is given sc on day of embryo transfer
  Other Names: prontogest 100 mg ampoles

SUMMARY:
Study if supporting luteal phase of high responder (high egg production or high Estradiol level) long Gn_Rh agonist protocol ICSI/IVF cycle by combined Estradiol and progesterone impairs or improves outcome in terms of pregnancy and implanation rates.

DETAILED DESCRIPTION:
The role of estradiol (E2) luteal support is still debated after more than a decade of use. Two recent met analyses (Gelbaya et al 2008) &(Jee et al 2010)( ) has shown that the addition of E2 to P4 for luteal phase support in IVF/ICSI cycles has no beneficial effect on pregnancy rates. However they commented that the data in the literature are, limited and heterogeneous, precluding the extraction of clear and definite conclusions. Previous met analysis ( Pritts and Atwood 2002 ) and an update (Fatemi et al 2007 ) and subsequent randomized trials ( Ghanem et al 2009 , Var et al 2011 ) reported beneficial effects of adding E2 to luteal P4 support. Recent retrospective studies have shown that high response in terms of excess egg production ( >15 . ) and or high E2 (Chen et al 2007,Kyrou et al 2009, Sunkara 2011 ) are detrimental to cycle outcome. This prospective randomized trial aims to study whether adding E2 to P4 luteal support in high ovarian responders is detrimental to cycle outcome or not

--------------- Gelbaya TA, KyrgiouM, Tsoumpou I, Nardo LG. The use of estradiol for luteal phase support in in vitro fertilization/intracytoplasmic sperminjec- tion cycles: a systematic review and meta-analysis. Fertil Steril 2008;90: 2116-25.

Jee BC, Suh CS, Kim SH, Kim YB, Moon SY. Effects of estradiol supplementation during the luteal phase of in vitro fertilization cycles: a meta-analysis Fertil Steril. 2010 Feb;93(2):428-36

Pritts EA, Atwood AK. Luteal phase support in infertility treatment: a meta-analysis of randomized trials. Hum Reprod 2002;17:2287-99 Fatemi HM, Popovic-Todorovic B, Papanikolaou E, Donoso P,Devroey P. An update of luteal phase support in stimulated IVF cycles.Hum Reprod Update 2007;13:581.

* Ghanem M E., Ehab E. Sadek, Elboghdady L. A.. Helal A S, Gamal Anas, Eldiasty A Bakre N I., Houssen M .The effect of luteal phase support protocol on cycle outcome and luteal phase hormone profile in long agonist protocol intracytoplasmic sperm injection cycles: a randomized clinical trial , Fertility and Sterility 2009 92: 486-493

Var T, Tonguc EA, Doğanay M, Gulerman C, Gungor T, Mollamahmutoglu L. A comparison of the effects of three different luteal phase support protocols on in vitro fertilization outcomes: a randomized clinical trial. Fertil Steril. 2011 Mar 1;95(3):985-9.

van der Gaast, Eijkemans JB, de Boer EJ, Burger CW , van Leeuwen FE, Fauser BCJM , and Macklon NS Optimum number of oocytes for a successful first IVF treatment cycle Reproductive BioMedicine Online 2006 ; 13: 476-480

Sunkara SK, Rittenberg V, Raine-Fenning N, Bhattacharya S, Zamora J, Coomarasamy A. Association between the number of eggs and live birth in IVF treatment: an analysis of 400 135 treatment cycles. Hum Reprod 2011; 26: 1768-1774

Chen QJ, Sun XX, Li L, Gao XH, Wu Y, Gemzell-Danielsson K, Cheng LN Effects of ovarian high response on implantation and pregnancy outcome during controlled ovarian hyperstimulation (with GnRH agonist and rFSH). Acta Obstet Gynecol Scand. 2007;86:849-54 Kyrou D., Popovic-Todorovic B., Fatemi H.M1, Bourgain C, Haentjens P., Van Landuyt L., and. Devroey P Does the estradiol level on the day of human chorionic gonadotrophin administration have an impact on pregnancy rates in patients treated with rec-FSH/GnRH antagonist? Hum Reprod 2009, 2902-2909,

ELIGIBILITY:
Inclusion criteria

* age<40 years,
* first ICSI cycle,
* third day FSH< 10 mIU/mL,
* serum E2 level on day of hCG administration <4,000 pg/mL,
* number of ova obtained >15

Exclusion Criteria:

* age 40 years or more,
* basal FSH 10 mIU/mL or more ,
* eggs retrieved 15 or less ,
* E2 level on day of hCG administration 4000 or more pg/ mL or more,
* repeat ICSI , need for PGD, presence of myoma , hydrosalpinx (unless disconnected)

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
cycle pregnancy rate | 6 weeks
  pregnancy rate per started cycle

SECONDARY OUTCOMES:
implantation rate, multiple pregnancy rate, ongoing pregnancy rate ,live birth rate | 6 weeks
  implantation rate,multible pregnancy rate, abortion rate

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura Integrated fertility center, Al Mansurah, Dekahlia, Egypt

REFERENCES:
- [Background] Gelbaya TA, Kyrgiou M, Tsoumpou I, Nardo LG. The use of estradiol for luteal phase support in in vitro fertilization/intracytoplasmic sperm injection cycles: a systematic review and meta-analysis. Fertil Steril. 2008 Dec;90(6):2116-25. doi: 10.1016/j.fertnstert.2007.10.053. Epub 2008 Jan 7. PMID 18178194
- [Background] Sunkara SK, Rittenberg V, Raine-Fenning N, Bhattacharya S, Zamora J, Coomarasamy A. Association between the number of eggs and live birth in IVF treatment: an analysis of 400 135 treatment cycles. Hum Reprod. 2011 Jul;26(7):1768-74. doi: 10.1093/humrep/der106. Epub 2011 May 10. PMID 21558332